CLINICAL TRIAL: NCT00078806
Title: A Phase 3 Safety and Efficacy Study of Etanercept In Children With Systemic Onset Juvenile Rheumatoid Arthritis
Brief Title: Safety and Efficacy Study of Etanercept (Enbrel®) In Children With Systemic Onset Juvenile Rheumatoid Arthritis
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: the study was terminated because of slow enrollment
Sponsor: Amgen (Industry)
Collaborators: Immunex Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 20021631; NCT00039949 (obsolete NCT alias)
Record Dates: First submitted 2004-03-05; First posted 2004-03-09 (Estimated); Results first posted 2019-09-25 (Actual); Last update posted 2019-09-25 (Actual); Status verified 2019-08

CONDITIONS: Juvenile Rheumatoid Arthritis
Keywords: Systemic Onset Juvenile Rheumatoid Arthritis; SOJRA; Fever; Rash; Joint Pain
MeSH Terms: conditions — Arthritis, Juvenile; Fever; Exanthema; Arthralgia | interventions — Etanercept

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (4):
- Part 1: Etanercept (Experimental): Participants received 0.4 mg/kg etanercept administered subcutaneously twice a week for up to 6 months in Part 1A.
  Participants who had a partial response entered Part 1B and received 0.8 mg/kg etanercept twice weekly for up to 4 months.
  Interventions: Drug: Etanercept
- Part 2: Placebo (Placebo Comparator): Participants who met response criteria in Part 1 were randomized to receive placebo twice a week for up to 3 months.
  Interventions: Drug: Placebo
- Part 2: Etanercept (Experimental): Participants who met response criteria in Part 1 were randomized to continue receiving etanercept twice a week at the same dose as in Part 1 (0.4 or 0.8 mg/kg) for up to 3 months.
  Interventions: Drug: Etanercept
- Part 3: (Experimental): Participants who experienced a flare or completed 3 months of treatment in Part 2 entered Part 3 and received open-label treatment with etanercept at the same dose as in Part 1 (0.4 or 0.8 mg/kg) for up to a maximum of 12 months, including treatment in Part 2.
  Interventions: Drug: Etanercept

INTERVENTIONS:
Drug: Etanercept — Administered by subcutaneous injection twice a week
  Other Names: Enbrel
  Arms: Part 1: Etanercept; Part 2: Etanercept; Part 3:
Drug: Placebo — Administered by subcutaneous injection twice a week
  Arms: Part 2: Placebo

SUMMARY:
The primary objective of this study was to determine the efficacy of etanercept in pediatric patients with systemically active system onset juvenile rheumatoid arthritis (SOJRA).

DETAILED DESCRIPTION:
Participants were to receive etanercept at a dose of 0.4 mg/kg twice weekly in Part 1A. Participants who had a partial response (not able to reduce prednisone dose by 50% of the baseline dose in 5 months) while on 0.4 mg/kg twice weekly etanercept in Part 1A were to enter Part 1B for up to 4 months and were to have the dose of etanercept increased to 0.8 mg/kg twice weekly. Participants who did not meet the response criteria in Part 1A or Part 1B of the study were to be withdrawn from the study as non-responders. Participants who responded in either Part 1A or Part 1B were randomized into Part 2, where they received etanercept or matching placebo in a double-blind manner twice weekly for up to 3 months. In Part 2, participants were stratified by the dosage of etanercept (0.4 mg/kg or 0.8 mg/kg) they were receiving in Part 1A or Part 1B. Participants could enter Part 3, the open-label re-treatment portion of the study, only if they had been entered into Part 2 of the study and had either flared in Part 2 or had completed 3 months of treatment in Part 2. The maximum time participants could receive etanercept in Part 2 and Part 3 combined was 12 months.

ELIGIBILITY:
INCLUSION CRITERIA:

* 2 - 18 years of age
* SOJRA for at least 3 months, with stable systemic features
* If taking methotrexate, hydroxychloroquine, or NSAIDs, dose must be stable
* Must take prednisone at a stable dose

EXCLUSION CRITERIA:

* Need for other DMARDs or prestudy requirements for oral or parenteral pulse steroids or intra-articular steroids
* Pregnant or nursing female
* Clinically significant abnormal laboratory test results for blood cells, liver or kidney function, or serology
* Previous receipt of any tumor necrosis factor (TNF) inhibitor
* Live virus vaccine within 12 weeks of study entry
* Participation in another study requiring informed consent within 12 weeks of entry
* Diabetes that requires insulin treatment
* Infection, chronic, recurrent, or currently active
* Any serious medical or psychiatric condition or history of alcohol or drug abuse

Ages: 2 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 19 (Actual)
Dates: Start 2001-06-04 (Actual); Primary Completion 2004-05-06 (Actual); Study Completion 2004-05-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: MD, Study Director — Amgen

REFERENCES:
- See also: AmgenTrials clinical trials website — http://www.amgentrials.com
- See also: Notice regarding posted summaries of trial results — http://download.veritasmedicine.com/REGFILES/amgen/Amgen_results_disclaimer.pdf
- See also: To access clinical trial results information click on this link — http://download.veritasmedicine.com/REGFILES/amgen/08D_FDAMA_113_Posting_Summary_916_ENBREL_20021631.pdf
- See also: FDA-approved Drug Labeling — http://www.enbrel.com/

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants with systemic onset juvenile rheumatoid arthritis (SOJRA) were enrolled at 7 sites in the United States and 4 sites in Canada.
Pre-assignment Details: Participants who responded in Part 1A or 1B were randomized into Part 2, stratified by the dosage of etanercept (0.4 mg/kg or 0.8 mg/kg) they received in Part 1. Participants entered Part 3 only if they had either flared in Part 2 or had completed 3 months of treatment in Part 2. Participants who did not respond in Part 1A or 1B were withdrawn.
Groups:
- Part 3: Etanercept: Participants who experienced a flare in Part 2 or completed 3 months of treatment in Part 2 entered Part 3 and received open-label treatment with etanercept at the same dose as in Part 1 (0.4 or 0.8 mg/kg) for up to a maximum of 12 months, including Part 2.
Period: Part 1A
Arm/Group | Part 1: Etanercept | Part 2: Placebo | Part 2: Etanercept | Part 3: Etanercept
Started | 19 | 0 | 0 | 0
Completed | 9 | 0 | 0 | 0
Not Completed | 10 | 0 | 0 | 0
Not completed — Adverse Event | 2 | 0 | 0 | 0
Not completed — Lack of Efficacy | 7 | 0 | 0 | 0
Not completed — Other | 1 | 0 | 0 | 0
Period: Part 1B
Arm/Group | Part 1: Etanercept | Part 2: Placebo | Part 2: Etanercept | Part 3: Etanercept
Started | 10 | 0 | 0 | 0
Completed | 2 | 0 | 0 | 0
Not Completed | 8 | 0 | 0 | 0
Not completed — Adverse Event | 1 | 0 | 0 | 0
Not completed — Lack of Efficacy | 7 | 0 | 0 | 0
Period: Part 2
Arm/Group | Part 1: Etanercept | Part 2: Placebo | Part 2: Etanercept | Part 3: Etanercept
Started | 0 | 6 | 4 | 0
Received Study Drug | 0 | 5 | 4 | 0
Completed | 0 | 5 | 4 | 0
Not Completed | 0 | 1 | 0 | 0
Not completed — Adverse Event | 0 | 1 | 0 | 0
Period: Part 3
Arm/Group | Part 1: Etanercept | Part 2: Placebo | Part 2: Etanercept | Part 3: Etanercept
Started | 0 | 0 | 0 | 9
Completed | 0 | 0 | 0 | 9
Not Completed | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: All enrolled participants
Arm/Group | Part 1: Etanercept
Number analyzed (Participants) | 19
Age, Continuous [Mean (Standard Deviation); unit: years] | 9.05 (4.20)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10
  Male | 9
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 15
  Hispanic | 2
  Other | 2

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants in Part 2 With Disease Flare
Description: Disease flare was defined as the presence of:
  * 1 major flare criterion plus 1 minor flare criterion or 1 lab criterion, OR
  * 2 minor flare criteria plus 2 lab criteria
  Major Criteria:
  * Fever of SOJRA, defined as a spike in axillary temperature ≥ 100°F (38°C) for ≥ 2 days per week in the prior 2 weeks or 8 days during the prior month
  * Symptomatic serositis documented by x-ray or other imaging modality Minor Flare Criteria
  * Rash of SOJRA, documented in the daily diary
  * Splenomegaly defined as spleen palpable > 2 cm below the left costal margin
  * Lymphadenopathy defined as ≥ 1 cm in > 1 node area
  * Arthritis defined as ≥ 2 active joints with swelling not due to deformity, or if swelling is absent, then 2 joints with loss of motion with pain on passive motion and/or warmth.
  Laboratory Criteria:
  All labs should be outside the normal range and with 30% worsening:
  * Albumin
  * Platelet count
  * Hemoglobin
  * C-reactive protein (CRP) or erythrocyte sedimentation rate (ESR)
Time Frame: 3 months during Part 2 (depending on the timing of response, entry into Part 2 was between study months 3 and 10)
Population: Participants randomized into Part 2 who received at least 1 dose of study drug in Part 2 (placebo or etanercept).
Measure: Count of Participants; unit: Participants
Arm/Group | Part 2: Placebo | Part 2: Etanercept
Number analyzed (Participants) | 5 | 4
Participants | 1 | 0

2. Secondary Outcome: Number of Participants With Adverse Events
Time Frame: Part 1A, maximum duration on treatment was 207 days; Part 1B, maximum duration on treatment was 120 days; Part 2, maximum duration on treatment was 88 days; Part 3, maximum duration on treatment was 130 days; plus 30 days after last dose of study drug.
Population: Participants who entered each part of the study and received study drug in each part of the study.
Measure: Count of Participants; unit: Participants
Groups:
- Part 1A: Etanercept 0.4 mg/kg: Participants received 0.4 mg/kg etanercept administered subcutaneously twice a week for up to 6 months in Part 1A.
- Part 1B: Etanercept 0.8 mg/kg: Participants in Part A1 who had a partial response entered Part 1B and received 0.8 mg/kg etanercept twice weekly for up to 4 months.
Arm/Group | Part 1A: Etanercept 0.4 mg/kg | Part 1B: Etanercept 0.8 mg/kg | Part 2: Placebo | Part 2: Etanercept | Part 3: Etanercept
Number analyzed (Participants) | 19 | 8 | 5 | 4 | 9
Participants
  Non-infectious adverse events | 16 | 3 | 2 | 2 | 4
  Infectious adverse events | 14 | 2 | 4 | 1 | 3

3. Secondary Outcome: Time to Flare in Part 2
Description: Time to flare was defined as the time from first dose of etanercept in Part 1 to the date of flare during Part 2.
Time Frame: From first dose in Part 1 to the end of Part 2 (up to 13 months)
Population: Participants randomized in Part 2 with a flare in Part 2
Measure: Median (Full Range); unit: days
Arm/Group | Part 2: Placebo | Part 2: Etanercept
Number analyzed (Participants) | 1 | 0
days | 180 [180 to 180] |

4. Secondary Outcome: Change From Baseline in Physician Global Assessment of Disease Severity in Part 1
Description: Physician global assessment of disease severity assessed on a visual analog scale (VAS) from 0 (asymptomatic) to 10 (severe symptoms).
Time Frame: Baseline and months 1, 2, 3, 4, 5, 6, 7, 8, and 9
Population: Participants who enrolled in the study and received at least one dose of etanercept in Part 1A or Part 1B and with available data at each time point.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Part 1: Etanercept
Number analyzed (Participants) | 19
units on a scale
  Month 1 | -1.42 (2.34)
  Month 2 | -2.21 (2.57)
  Month 3 | -1.26 (2.62)
  Month 4: number analyzed (Participants) | 17
  Month 4 | -1.82 (2.53)
  Month 5: number analyzed (Participants) | 15
  Month 5 | -2.13 (2.36)
  Month 6: number analyzed (Participants) | 11
  Month 6 | -1.64 (2.58)
  Month 7: number analyzed (Participants) | 5
  Month 7 | -0.40 (1.82)
  Month 8: number analyzed (Participants) | 2
  Month 8 | 0.50 (2.12)
  Month 9: number analyzed (Participants) | 2
  Month 9 | 0.00 (1.41)

5. Secondary Outcome: Change From Baseline in Physician Global Assessment of Disease Severity in Part 2
Description: as for outcome 4
Time Frame: Baseline and months 5, 6, 7, 8, and 9
Population: Participants who randomized and received at least one dose of study drug in Part 2 and with available data at each time point; participants could join Part 2 at different times depending on their response status.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Part 2: Placebo | Part 2: Etanercept
Number analyzed (Participants) | 5 | 4
units on a scale
  Month 5: number analyzed (Participants) | 1 | 1
  Month 5 | -1.00 (NA) — Could not be calculated for N=1 | -4.00 (NA) — Could not be calculated for N=1
  Month 6: number analyzed (Participants) | 2 | 2
  Month 6 | -0.50 (2.12) | -3.00 (1.41)
  Month 7: number analyzed (Participants) | 3 | 4
  Month 7 | -3.67 (1.53) | -4.25 (0.50)
  Month 8: number analyzed (Participants) | 4 | 3
  Month 8 | -4.00 (1.83) | -2.67 (2.52)
  Month 9: number analyzed (Participants) | 3 | 1
  Month 9 | -4.67 (1.53) | -6.00 (NA) — Could not be calculated for N=1

6. Secondary Outcome: Change From Baseline in Patient's/Parent's Global Assessment in Part 1
Description: Patient's/parent's global assessment of overall well-being assessed on a visual analog scale (VAS) from 0 (asymptomatic) to 10 (severe symptoms).
Time Frame: Baseline and months 1, 2, 3, 4, 5, 6, 7, 8, and 9
Population: Participants who enrolled in the study and received at least one dose of etanercept in Part 1A or Part 1B and with available data at baseline and each time point.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Part 1: Etanercept
Number analyzed (Participants) | 18
units on a scale
  Month 1: number analyzed (Participants) | 17
  Month 1 | -1.88 (2.52)
  Month 2: number analyzed (Participants) | 16
  Month 2 | -2.38 (2.63)
  Month 3: number analyzed (Participants) | 16
  Month 3 | -1.44 (3.46)
  Month 4: number analyzed (Participants) | 14
  Month 4 | -2.50 (2.62)
  Month 5: number analyzed (Participants) | 13
  Month 5 | -2.54 (2.93)
  Month 6: number analyzed (Participants) | 9
  Month 6 | -2.89 (2.09)
  Month 7: number analyzed (Participants) | 5
  Month 7 | -2.00 (3.32)
  Month 8: number analyzed (Participants) | 2
  Month 8 | -0.50 (0.71)
  Month 9: number analyzed (Participants) | 1
  Month 9 | 0.00 (NA) — Could not be calculated when N=1

7. Secondary Outcome: Change From Baseline in Patient's/Parent's Global Assessment of Disease Severity in Part 2
Description: as for outcome 6
Time Frame: Baseline and months 5, 6, 7, 8, and 9
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Part 2: Placebo | Part 2: Etanercept
Number analyzed (Participants) | 5 | 4
units on a scale
  Month 5: number analyzed (Participants) | 1 | 1
  Month 5 | 0.00 (NA) — Cannot be calculated when N=1 | -7.00 (NA) — Cannot be calculated when N=1
  Month 6: number analyzed (Participants) | 2 | 2
  Month 6 | -3.00 (4.24) | -5.00 (2.83)
  Month 7: number analyzed (Participants) | 3 | 4
  Month 7 | -3.33 (0.58) | -4.25 (1.89)
  Month 8: number analyzed (Participants) | 4 | 3
  Month 8 | -4.25 (2.22) | -2.67 (2.31)
  Month 9: number analyzed (Participants) | 3 | 1
  Month 9 | -5.33 (0.58) | -5.00 (NA) — Cannot be calculated when N=1

8. Secondary Outcome: Change From Baseline in Number of Active Joints in Part 1
Description: Active joints are those with swelling not due to bony deformity or if swelling is absent, loss of motion (LOM) accompanied by pain on passive motion and/or tenderness and/or warmth.
Time Frame: Baseline and months 1, 2, 3, 4, 5, 6, 7, 8, and 9
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: active joints
Arm/Group | Part 1: Etanercept
Number analyzed (Participants) | 18
active joints
  Month 1: number analyzed (Participants) | 17
  Month 1 | -1.94 (6.65)
  Month 2: number analyzed (Participants) | 16
  Month 2 | -6.75 (10.35)
  Month 3: number analyzed (Participants) | 16
  Month 3 | -3.50 (18.89)
  Month 4: number analyzed (Participants) | 14
  Month 4 | -3.21 (5.42)
  Month 5: number analyzed (Participants) | 13
  Month 5 | -5.46 (9.20)
  Month 6: number analyzed (Participants) | 11
  Month 6 | -1.55 (8.72)
  Month 7: number analyzed (Participants) | 6
  Month 7 | -1.83 (5.19)
  Month 8: number analyzed (Participants) | 3
  Month 8 | -1.67 (8.08)
  Month 9: number analyzed (Participants) | 2
  Month 9 | -4.00 (4.24)

9. Secondary Outcome: Change From Baseline in Number of Active Joints in Part 2
Description: as for outcome 8
Time Frame: Baseline and months 5, 6, 7, 8, and 9
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: active joints
Arm/Group | Part 2: Placebo | Part 2: Etanercept
Number analyzed (Participants) | 5 | 4
active joints
  Month 5: number analyzed (Participants) | 1 | 0
  Month 5 | -12.00 (NA) — Could not be calculated when N=1 |
  Month 6: number analyzed (Participants) | 2 | 2
  Month 6 | -11.50 (7.78) | -11.00 (12.73)
  Month 7: number analyzed (Participants) | 3 | 2
  Month 7 | -6.33 (4.51) | -17.00 (9.90)
  Month 8: number analyzed (Participants) | 3 | 3
  Month 8 | -4.67 (2.08) | -13.00 (5.00)
  Month 9: number analyzed (Participants) | 1 | 0
  Month 9 | -25.00 (NA) — Cannot be calculated when N=1 |

10. Secondary Outcome: Change From Baseline in Number of Joints With Limitation of Motion in Part 1
Time Frame: Baseline and months 1, 2, 3, 4, 5, 6, 7, 8, and 9
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: joints
Arm/Group | Part 1: Etanercept
Number analyzed (Participants) | 18
joints
  Month 1 | 0.50 (7.34)
  Month 2: number analyzed (Participants) | 16
  Month 2 | -0.19 (6.49)
  Month 3: number analyzed (Participants) | 17
  Month 3 | 1.88 (15.11)
  Month 4: number analyzed (Participants) | 15
  Month 4 | 1.27 (7.71)
  Month 5: number analyzed (Participants) | 12
  Month 5 | -0.92 (3.78)
  Month 6: number analyzed (Participants) | 9
  Month 6 | 2.56 (7.06)
  Month 7: number analyzed (Participants) | 5
  Month 7 | -0.40 (6.15)
  Month 8: number analyzed (Participants) | 3
  Month 8 | -1.33 (7.64)
  Month 9: number analyzed (Participants) | 2
  Month 9 | -5.50 (6.36)

11. Secondary Outcome: Change From Baseline in Number of Joints With Limitation of Motion in Part 2
Time Frame: Baseline and months 5, 6, 7, 8, and 9
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: joints
Arm/Group | Part 2: Placebo | Part 2: Etanercept
Number analyzed (Participants) | 5 | 4
joints
  Month 5: number analyzed (Participants) | 1 | 1
  Month 5 | 4.0 (NA) — Could not be calculated when N=1 | -2.00 (NA) — Could not be calculated when N=1
  Month 6: number analyzed (Participants) | 2 | 1
  Month 6 | 4.50 (2.12) | 26.00 (NA) — Could not be calculated when N=1
  Month 7: number analyzed (Participants) | 3 | 4
  Month 7 | 2.67 (4.73) | -3.00 (5.94)
  Month 8: number analyzed (Participants) | 4 | 3
  Month 8 | 1.75 (4.86) | 1.00 (8.19)
  Month 9: number analyzed (Participants) | 3 | 0
  Month 9 | -8.00 (13.89) |

12. Secondary Outcome: Change From Baseline in Childhood Health Assessment Questionnaire (CHAQ) Disability Index in Part 1
Description: Childhood Health Assessment Questionnaire (CHAQ) disability index is used to assess physical functioning in children with arthritis. The scale consists of 30 questions in 8 domains (dressing, grooming, arising, eating, walking, reach, grip, and activities). Each question is scored on a scale from 0 to 3, where 0 = Without any difficulty; 1 = With some difficulty; 2 = With much difficulty; 3 = Unable to do. The overall score ranges from 0 (no difficulty) to 3 (unable to do).
Time Frame: Baseline and months 1, 2, 3, 4, 5, 6, 7, 8, and 9
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Part 1: Etanercept
Number analyzed (Participants) | 19
units on a scale
  Month 1 | -0.35 (0.74)
  Month 2 | -0.30 (0.68)
  Month 3 | -0.27 (0.72)
  Month 4: number analyzed (Participants) | 16
  Month 4 | -0.29 (0.73)
  Month 5: number analyzed (Participants) | 14
  Month 5 | -0.47 (0.84)
  Month 6: number analyzed (Participants) | 9
  Month 6 | -0.57 (1.15)
  Month 7: number analyzed (Participants) | 6
  Month 7 | -0.29 (0.66)
  Month 8: number analyzed (Participants) | 2
  Month 8 | -0.06 (1.50)
  Month 9: number analyzed (Participants) | 2
  Month 9 | 0.25 (1.06)

13. Secondary Outcome: Change From Baseline in Childhood Health Assessment Questionnaire (CHAQ) Disability Index in Part 2
Description: as for outcome 12
Time Frame: Baseline and months 5, 6, 7, 8, and 9
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Part 2: Placebo | Part 2: Etanercept
Number analyzed (Participants) | 5 | 4
units on a scale
  Month 5: number analyzed (Participants) | 1 | 1
  Month 5 | 0.0 (NA) — Could not be calculated when N=1 | -1.63 (NA) — Could not be calculated when N=1
  Month 6: number analyzed (Participants) | 2 | 2
  Month 6 | -0.06 (0.09) | -0.75 (1.24)
  Month 7: number analyzed (Participants) | 3 | 4
  Month 7 | -1.08 (1.23) | -0.63 (1.18)
  Month 8: number analyzed (Participants) | 4 | 3
  Month 8 | -1.09 (1.19) | -0.29 (0.56)
  Month 9: number analyzed (Participants) | 3 | 1
  Month 9 | -1.54 (1.44) | -1.50 (NA) — Could not be calculated when N=1

14. Secondary Outcome: Change From Baseline in C-reactive Protein (CRP) Levels in Part 1
Time Frame: Baseline and months 1, 2, 3, 4, 5, 6, 7, 8, and 9
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Part 1: Etanercept
Number analyzed (Participants) | 6
mg/dL
  Month 1: number analyzed (Participants) | 5
  Month 1 | -4.13 (6.10)
  Month 2: number analyzed (Participants) | 5
  Month 2 | -4.23 (9.53)
  Month 3: number analyzed (Participants) | 5
  Month 3 | -4.04 (6.80)
  Month 4: number analyzed (Participants) | 4
  Month 4 | -6.03 (7.66)
  Month 5: number analyzed (Participants) | 2
  Month 5 | -3.07 (3.71)
  Month 6: number analyzed (Participants) | 1
  Month 6 | -5.97 (NA) — Could not be calculated when N=1
  Month 7: number analyzed (Participants) | 0
  Month 8: number analyzed (Participants) | 0
  Month 9: number analyzed (Participants) | 0

15. Secondary Outcome: Change From Baseline in C-reactive Protein (CRP) Levels in Part 2
Time Frame: Baseline and months 5, 6, 7, 8, and 9
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Part 2: Placebo | Part 2: Etanercept
Number analyzed (Participants) | 5 | 4
mg/dL
  Month 5: number analyzed (Participants) | 1 | 0
  Month 5 | -0.44 (NA) — Could not be calculated when N=1 |
  Month 6: number analyzed (Participants) | 1 | 1
  Month 6 | 1.88 (NA) — Could not be calculated when N=1 | -0.77 (NA) — Could not be calculated when N=1
  Month 7: number analyzed (Participants) | 0 | 2
  Month 7 |  | -3.43 (3.60)
  Month 8: number analyzed (Participants) | 0 | 2
  Month 8 |  | -3.43 (3.60)
  Month 9: number analyzed (Participants) | 0 | 1
  Month 9 |  | -5.97 (NA) — Could not be calculated when N=1

ADVERSE EVENTS:
Time Frame: Part 1A, maximum duration on treatment was 207 days. Part 1B, maximum duration on treatment was 120 days Part 2, maximum duration on treatment was 88 days Part 3, maximum duration on treatment was 130 days Plus one month after the last dose of study drug.
Description: Other Adverse Events summarizes the non-serious occurrences of adverse events that exceed the indicated frequency threshold.
Groups:
- Part 1B: Etanercept 0.8 mg/kg: Participants who had a partial response in Part 1A entered Part 1B and received 0.8 mg/kg etanercept twice weekly for up to 4 months.
- Part 2: Placebo: Participants who met response criteria in Part 1 were randomized to receive placebo twice a week for up to 3 months in Part 2.
- Part 2: Etanercept 0.4/0.8 mg/kg: Participants who met response criteria in Part 1 were randomized to continue receiving etanercept twice a week at the same dose as in Part 1 (0.4 or 0.8 mg/kg) for up to 3 months in Part 2.
- Part 3: Etanercept 0.4/0.8 mg/kg: Participants who experienced a flare or completed 3 months of treatment in Part 2 entered Part 3 and received open-label treatment with etanercept at the same dose as in Part 1 (0.4 or 0.8 mg/kg) for up to a maximum of 12 months, including treatment received in Part 2.
Arm/Group | Part 1A: Etanercept 0.4 mg/kg | Part 1B: Etanercept 0.8 mg/kg | Part 2: Placebo | Part 2: Etanercept 0.4/0.8 mg/kg | Part 3: Etanercept 0.4/0.8 mg/kg
Serious Adverse Events (participants affected / at risk) | 3/19 | 1/8 | 0/5 | 0/4 | 0/9
Other Adverse Events (participants affected / at risk) | 18/19 | 4/8 | 4/5 | 3/4 | 5/9
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Part 1A: Etanercept 0.4 mg/kg (N=19) | Part 1B: Etanercept 0.8 mg/kg (N=8) | Part 2: Placebo (N=5) | Part 2: Etanercept 0.4/0.8 mg/kg (N=4) | Part 3: Etanercept 0.4/0.8 mg/kg (N=9)
Anaemia (Blood and lymphatic system disorders) | 1 | 0 | 0 | 0 | 0
Gastroenteritis (Infections and infestations) | 1 | 0 | 0 | 0 | 0
Rheumatoid arthritis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0
Pleurisy (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Part 1A: Etanercept 0.4 mg/kg (N=19) | Part 1B: Etanercept 0.8 mg/kg (N=8) | Part 2: Placebo (N=5) | Part 2: Etanercept 0.4/0.8 mg/kg (N=4) | Part 3: Etanercept 0.4/0.8 mg/kg (N=9)
Anaemia (Blood and lymphatic system disorders) | 1 | 0 | 0 | 0 | 0
Ear pain (Ear and labyrinth disorders) | 1 | 0 | 0 | 0 | 0
Cataract (Eye disorders) | 1 | 0 | 0 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 2 | 0 | 0 | 0 | 0
Abdominal pain upper (Gastrointestinal disorders) | 3 | 0 | 0 | 0 | 0
Aphthous ulcer (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 1
Cheilosis (Gastrointestinal disorders) | 1 | 0 | 1 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 2 | 0 | 0 | 1 | 0
Nausea (Gastrointestinal disorders) | 2 | 0 | 0 | 0 | 0
Vomiting (Gastrointestinal disorders) | 2 | 0 | 0 | 0 | 0
Fatigue (General disorders) | 2 | 0 | 0 | 0 | 0
Feeling hot (General disorders) | 1 | 0 | 0 | 0 | 0
Injection site bruising (General disorders) | 1 | 0 | 0 | 0 | 0
Injection site erythema (General disorders) | 3 | 0 | 0 | 0 | 0
Injection site pruritus (General disorders) | 3 | 0 | 0 | 0 | 0
Injection site rash (General disorders) | 1 | 0 | 1 | 0 | 0
Injection site reaction (General disorders) | 7 | 0 | 0 | 1 | 2
Drug hypersensitivity (Immune system disorders) | 2 | 0 | 0 | 0 | 0
Bronchitis (Infections and infestations) | 1 | 0 | 0 | 0 | 0
Conjunctivitis (Infections and infestations) | 0 | 0 | 0 | 0 | 1
Epstein-Barr viraemia (Infections and infestations) | 0 | 1 | 0 | 0 | 0
Herpes simplex (Infections and infestations) | 1 | 0 | 0 | 0 | 0
Herpes zoster (Infections and infestations) | 1 | 0 | 0 | 0 | 0
Influenza (Infections and infestations) | 0 | 0 | 0 | 0 | 1
Nasopharyngitis (Infections and infestations) | 0 | 0 | 0 | 1 | 0
Oral herpes (Infections and infestations) | 1 | 0 | 0 | 0 | 0
Otitis media (Infections and infestations) | 1 | 0 | 1 | 0 | 0
Paronychia (Infections and infestations) | 1 | 0 | 0 | 0 | 0
Pharyngitis (Infections and infestations) | 1 | 0 | 1 | 0 | 0
Pharyngitis streptococcal (Infections and infestations) | 2 | 0 | 0 | 0 | 0
Sinusitis (Infections and infestations) | 1 | 0 | 0 | 0 | 0
Upper respiratory tract infection (Infections and infestations) | 6 | 2 | 2 | 0 | 2
Urinary tract infection (Infections and infestations) | 1 | 0 | 0 | 0 | 0
Viral infection (Infections and infestations) | 1 | 0 | 0 | 0 | 0
Fall (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0
Spinal fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0
Thermal burn (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0
Tooth injury (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1
Haemoglobin decreased (Investigations) | 0 | 0 | 0 | 0 | 1
Arthritis (Musculoskeletal and connective tissue disorders) | 2 | 0 | 0 | 0 | 0
Costochondritis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0
Flank pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0
Osteopenia (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0
Rheumatoid arthritis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0
Skin papilloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0 | 0
Dizziness (Nervous system disorders) | 2 | 0 | 0 | 0 | 0
Headache (Nervous system disorders) | 6 | 0 | 1 | 0 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 0 | 0 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0
Purpura (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1
Skin lesion (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Clinical Trial Agreement generally does not restrict an investigator's discussion of trial results after completion. The Agreement permits Amgen a limited period of time to review material discussing trial results (typically up to 45 days and possible extension). Amgen may remove confidential information, but authors have final control and approval of publication content. For multicenter studies, the investigator agrees not to publish any results before the first multi-center publication.